CLINICAL TRIAL: NCT07208994
Title: Pathways to Equitable Access to Kidney Transplantation in Spain (PATH2KT): A Transformative Mixed-methods Study Protocol
Brief Title: Pathways to Equitable Access to Kidney Transplantation in Spain: A Transformative Mixed-methods Study Protocol
Acronym: PATH2KT
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital del Mar (Other)
Collaborators: Organización Nacional de Trasplantes (ONT) (Unknown)
Responsible Party: Principal Investigator, GUILLERMO PEDREIRA ROBLES, Principal Investigator, Hospital del Mar
Other Study IDs: Hospital del Mar
Record Dates: First submitted 2025-06-27; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease; Kidney Transplant
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Description — No intervention

SUMMARY:
Introduction. Chronic kidney disease (CKD) affects 10%-15% of the global population and is projected to become the fifth leading cause of years of life lost by 2040. Despite the benefits of kidney transplantation (KT), access remains inequitable. In Spain, which leads the world in KT rates per million population, disparities may persist due to structural, territorial, and professional barriers. This study aims to explore the mechanisms underlying treatment deprivation and inequity in KT access using a mixed-methods approach.

Methods and analysis. A transformative mixed-methods design will be implemented in four phases: (1) systematic reviews on instruments assessing treatment deprivation and inequalities in CKD and KT; (2) a multicenter quantitative study and qualitative interviews with professionals and patients; (3) a pre-experimental evaluation of a training program on KT; and (4) triangulation and translation of findings to inform national policy. The protocol adheres to GRAMMS and PRISMA guidelines.

Ethics and dissemination. Approved by the Hospital del Mar Research Institute Ethics Committee (ID: XX), the study complies with EU data protection laws. Informed consent will be obtained. Findings will be disseminated via peer-reviewed publications, conferences, social media, and patient forums to support equity-focused strategies in KT.

DETAILED DESCRIPTION:
METHODS AND ANALYSIS >> Study design The design of this research protocol follows the premises of the mixed-methods approach under the transformative paradigm 26,27. This means that various phases of data collection -both quantitative and qualitative- will be conducted, analyzed separately, and then integrated through methodological triangulation to corroborate and enrich the findings 28. The research will be centered on social justice, amplifying the voices of communities facing health inequalities or treatment deprivation. Using the transformative mixed-methods approach, different power structures that may be involved in the results will be analyzed and linked to actions that promote equity, ultimately providing a report with recommendations for action based on the results obtained 26,27. The achievement of results under this methodology and paradigm will be accomplished through various research phases, explained in detail below.

This protocol follows the Good Reporting of A Mixed Methods Study (GRAMMS) guidelines, recognized for ensuring high-quality evidence-based methodology 29.

* Patient and public involvement This protocol has been reviewed and endorsed by the CKD community in Spain, including the National Federation of Associations for the Fight Against Kidney Diseases (ALCER) and the ADER Foundation (Kidney Patients Association of Catalonia). These organizations will actively support the dissemination of the study in different regions and will facilitate recruitment of participants during the data collection phase. Moreover, patient representatives will be involved in the interpretation of findings, ensuring that the analysis incorporates lived experiences and enhances the relevance and clarity of results.
* Study setting and context The data collection components of this research protocol will be conducted in Spain, a high-interest setting for the care of people with CKD. Spain's healthcare system is public and universal, primarily funded through taxes, ensuring healthcare access for the entire population, including individuals requiring KT 30. The country is internationally recognized for its high rates of organ donation and transplantation, supported by the Spanish National Transplant Organization (Organización Nacional de Trasplantes, ONT), which emphasizes coordination, regulation, and public engagement 31. Spain's healthcare system is also highly decentralized, with responsibilities for healthcare planning, service delivery, and resource allocation delegated to the 17 autonomous regions. This structure includes regional transplant coordination offices that work in alignment with the ONT to implement national policies at the local level, but may also reflect regional specificities and priorities. Despite this strong institutional framework, inequities in KT access might arise from factors such as socioeconomic status, geographic area and interregional differences linked to the decentralized organization of the healthcare system. By focusing solely on the Spanish context, while allowing for international discussion across the proposed phases, this study seeks to generate detailed insights and propose actionable recommendations grounded in the realities of Spain's healthcare infrastructure and sociopolitical landscape.
* Data collection and analysis Data collection and analysis will be carried out using a mixed approach, combining both quantitative and qualitative methods. This will result in four distinct research phases, tailored to the specific objectives of this research protocol.

  * Phase 1. Literature review The first phase of this study aims to address objectives 1 and 2, which focus on synthesizing and critically appraising the existing literature on instruments and variables used to evaluate inequities among individuals with CKD, as well as on examining how unequal access to KT is described and explained. To achieve this, two systematic reviews will be conducted.

Both reviews will be carried out following the methodological recommendations of the Joanna Briggs Institute (JBI) and will be reported according to the PRISMA 2020 guidelines 32,33. The protocols for the reviews will be registered in PROSPERO®. Searches will be conducted in the major electronic databases, using controlled vocabulary (MeSH) and will include peer-reviewed studies published between 2015 and 2025 in English, Spanish, French, or Portuguese. Eligibility criteria will be based on the PICOT framework, and include quantitative, qualitative, and mixed-methods research, as well as systematic and scoping reviews. Study selection, data extraction, and critical appraisal will be carried out independently by two or more reviewers, with discrepancies resolved by consensus or consultation with a third reviewer. Covidence® software will be used to manage the workflow.

Given the expected methodological heterogeneity, results will be synthesized narratively and organized thematically, according to the domains assessed, levels of analysis, validation approaches, and applicability of the instruments in both clinical and research contexts. These findings will provide a foundational knowledge base for the subsequent phases of the study.

> Phase 2. Inequities analysis This phase addresses objectives 3 and 4 by examining inequities in access to KT among individuals with CKD.

For the quantitative component (objective 3), a descriptive study will be conducted across Spain using a snowball sampling strategy through healthcare networks and patient organizations to ensure representativeness and inclusivity. Recruitment will continue until data saturation is reached, with a minimum of 500 participants to guarantee diversity across sociodemographic groups. Data will be collected through the questionnaires developed in Phase 1 (Appendix 1), complemented with sociodemographic and clinical variables to provide a comprehensive understanding of participants' health status and backgrounds. A multi-channel strategy will be applied to facilitate recruitment, involving healthcare professionals at nephrology and transplant centers, national and regional patient associations such as ALCER and ADER, and an online standardized interest form disseminated through institutional and collaborative networks, including ONT, SEDEN, and SEN. All participants will receive an information sheet and will be able to contact the research team directly to confirm their participation. No clinical information will be accessed without explicit consent, and contact details will only be shared if the participant initiates communication. This decentralized approach ensures voluntary participation and strict compliance with ethical standards in research involving potentially vulnerable populations. Statistical analysis will be carried out using SPSS® software. Descriptive statistics, including means, medians, standard deviations, and frequencies, will be used to summarize the sample characteristics, while inferential analyses such as t-tests, Wilcoxon tests, chi-square tests, and regression models will be applied depending on the type and distribution of the data. Assumptions for parametric tests will be verified, with non-parametric alternatives used when appropriate. Missing data will be managed through multiple imputation or complete-case analysis, depending on the extent and pattern of missingness, in order to ensure the robustness and validity of the findings.

For the qualitative component (objective 4), a descriptive study with a phenomenological orientation will be conducted to explore and understand in depth the experiences, perceptions, and meanings attributed to treatment deprivation by both healthcare professionals and individuals living with CKD. This approach will enable the identification of common patterns and differences between perspectives, providing a comprehensive view of the phenomenon from both sides of the healthcare relationship. Data will be collected through semi-structured, in-depth interviews guided by open-ended, non-directive questions designed to foster a fluid dialogue between interviewer and participant (Appendix 2). Two main groups of participants will be included: healthcare professionals involved in CKD care and KT, and patients with direct experience in the transplant process, including evaluation, waiting list, or transplantation. Healthcare professionals must have at least two years of experience in nephrology, transplant coordination, or related fields. Participants will be selected using purposive sampling with maximum variation to ensure diversity in roles, stages of CKD, and geographic regions. Interviews will be conducted by trained researchers or research assistants experienced in qualitative interviewing and working with vulnerable populations. Sessions will take place either in private spaces at participating healthcare centers (e.g., hospitals, transplant units, nursing schools) or through secure video calls, according to participants' preferences and availability, ensuring accessibility. Each interview is expected to last between 45 and 60 minutes, will be audio-recorded with prior consent, and subsequently transcribed verbatim for analysis. Follow-up interviews will be scheduled if necessary. Recruitment will continue until theoretical saturation is reached, defined as the point where no new themes or categories emerge from additional data 34. Data will be analyzed inductively using a thematic approach and content analysis to identify and categorize recurring patterns, with successive steps of coding, grouping into categories, and synthesizing into central themes. To ensure credibility and rigor, strategies such as investigator triangulation, participant validation, and reflective journaling of analytical decisions will be applied 35. All data will be anonymized using unique codes, stored securely, and handled in compliance with ethical standards. Atlas.ti software will be used to support the analytic process.

Upon completing this second research phase, we will have detailed data on inequities in access to KT in the Spanish context, together with the meanings attributed to this phenomenon by both the professional community and patients, providing comprehensive insights to inform the subsequent phases of the study.

> Phase 3. Impact of training In this third phase, objective 5 will be addressed by evaluating the impact of a training course in Spain on living donor KT for healthcare professionals. This particular course has been selected due to its established relevance within the Spanish context and potential impact upon access to KT: it has already completed three successful editions and has gained national recognition as one of the most important and well-regarded training programs on KT in Spain. Notably, the course is aimed at professionals working in non-transplant centers, particularly dialysis units and advanced CKD clinics, which positions it to directly influence early referral pathways and improve access to KT. Its consolidated presence and perceived influence on clinical practice make it a strategic candidate for evaluation.

A preexperimental quantitative study will be conducted with a pretest-posttest design. The study population will consist of healthcare professionals participating in the training, selected through convenience sampling. Data collection will be carried out through a structured questionnaire that will measure participants' knowledge, attitudes, and practices before, after, and one year after the course (Appendix 3). The questionnaire will include multiple-choice questions to assess knowledge, Likert scales to analyze attitudes, and questions about behaviors and clinical decision-making regarding living donor KT. The instrument's validity and reliability will be verified through prior piloting and consensus among the research team. Data analysis will involve descriptive statistics to characterize the sample and compare pre- and post-intervention results. Statistical tests such as the paired t-test or the Wilcoxon test, depending on the data distribution, will be applied to determine whether significant differences exist after training. Additionally, effect size measures, such as Cohen's d for continuous variables and Cramer's V for categorical variables, will be calculated to quantify the impact of the course on the evaluated variables.

The results obtained will help identify the effectiveness of the course in improving healthcare professionals' knowledge and perceptions about living donor KT, which can serve as the basis for future training strategies and for optimizing equitable access to KT within Spain.

> Phase 4. Integration of findings and contribution to the ATRAE national plan In the fourth and final phase of the project, the results obtained in the previous stages will be triangulated and synthesized to generate comprehensive, evidence-based knowledge (objective 6). This phase is conceived as an integrative component that will enable the transfer of research findings into actionable recommendations, directly contributing to the development of the national strategy for improving access to KT in Spain. The synthesis will support the creation of a consensus document within the ATRAE project: Optimizing Access to Kidney Transplantation in Spain. ATRAE is a national initiative led by the ONT, the Transplant Commission of the Interterritorial Council of the Spanish National Health System (CIT-SNS), and the Spanish Society of Nephrology (SEN), in collaboration with the Spanish Association of Urology (AEU), the Spanish Society of Nephrology Nursing (SEDEN), the Spanish Society of Immunology (SEI), and the Spanish Transplant Society (SET), and with the participation of the National Federation of Associations for the Fight Against Kidney Diseases (ALCER).

The research team will analyze and interpret the findings from both the quantitative and qualitative components, applying a triangulation process to enhance the validity and depth of interpretation. The results will be structured around key thematic areas such as regional disparities, evaluation and KT access processes, healthcare professional training, and the influence of social and structural determinants. Based on this synthesis, technical briefs will be prepared to highlight the most relevant insights, propose improvement strategies, and identify aspects that require further attention. These materials will be shared with the ATRAE working groups and coordination bodies, with the goal of supporting evidence-based decision-making and facilitating the integration of research findings into ongoing national planning processes.

Through this knowledge translation effort, the study positions itself as a relevant and timely contributor to the development of public policies, ensuring that its findings are not only scientifically rigorous but also transferable, actionable, and aligned with the institutional framework responsible for promoting equity in access to KT in Spain.

ELIGIBILITY:
Inclusion Criteria:

* People with CKD

Exclusion Criteria:

* Pediatrics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A transformative mixed-methods design will be implemented in four phases: (1) systematic reviews on instruments assessing treatment deprivation and inequalities in CKD and KT; (2) a multicenter quantitative study and qualitative interviews with professionals and patients; (3) a pre-experimental evaluation of a training program on KT; and (4) triangulation and translation of findings to inform national policy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Inequities in access to kidney transplantation among individuals with chronic kidney disease | Baseline (at study inclusion)
  Quantitative assessment of inequities in access to kidney transplantation using validated questionnaires developed in Phase 1, complemented by sociodemographic and clinical variables. The outcome will measure disparities according to age, sex, socioeconomic status, region, and clinical condition.

SECONDARY OUTCOMES:
Patient experiences related to access to kidney transplantation | Baseline (at study inclusion)
  Analysis of experiences collected through structured questionnaires to evaluate patients' perceptions of their health status, quality of life, and barriers or facilitators in the transplant process.
Professional perspectives on inequities in access to kidney transplantation | Within the first 12 months of the study
  Qualitative assessment through semi-structured interviews with nephrologists, nurses, healthcare managers, and patient advocates to explore their perceptions of systemic inequities and barriers in the transplant pathway.

OTHER OUTCOMES:
Thematic categories of inequities in kidney transplantation access | At study completion (24 months)
  Inductive thematic analysis of qualitative data to identify key categories and central themes related to inequities in transplantation access, triangulated with quantitative findings.

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Sanclemente Dalmau, Dr, Principal Investigator — Escola Superior d'Infermeria Hospital del Mar; Laura Rota Musoll, Dr, Principal Investigator — Universitat de Vic
Locations (1):
- Escola Superior d'Infermeria Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The following individual participant data (IPD) will be shared: de-identified sociodemographic variables (e.g., age, sex, region), clinical variables related to kidney disease stage and treatment modality, and responses to patient-reported outcome and experience measures (PROMs and PREMs) collected through standardized questionnaires. Data will be shared in aggregated and anonymized format to ensure confidentiality and will be used exclusively for research purposes in accordance with ethical approvals and participant consent.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) will become available after completion of the study and publication of the main results. Data will remain accessible for a period of 5 years following publication.
Access Criteria: De-identified individual participant data will be made available to qualified researchers upon reasonable request. Access will require submission of a research proposal that aligns with the study objectives, approval by the principal investigator, and a signed data access agreement to ensure compliance with ethical and legal standards.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT07208994/Prot_SAP_000.pdf